CLINICAL TRIAL: NCT02831699
Title: The Evaluation of Potential Zika, Chikungunya, and Dengue Infections in Mexico (Zik01)
Brief Title: The Evaluation of Potential Zika, Chikungunya, and Dengue Infections in Mexico
Acronym: Zik01
Status: Completed | Type: Observational
Sponsor: Mexican Emerging Infectious Diseases Clinical Research Network (Network)
Collaborators: Secretaria de Salud, Mexico (Other Government); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: Zik01
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Zika Virus Disease (Disorder); Dengue; Chikungunya
Keywords: Zika; Guillain Barré
MeSH Terms: conditions — Zika Virus Infection; Dengue; Chikungunya Fever; Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Febrile Rash
- Household
- Guillain-Barré prospective
- Prior Guillain-Barré

SUMMARY:
This study will evaluate subjects with fever and/or rash to determine the percentage of those infected by the Zika, Chikungunya, or Dengue virus. The study will also compare the clinical signs, symptoms, and lab abnormalities related to each virus, to better specify each virus's characteristics.

DETAILED DESCRIPTION:
The study will enroll subjects in several different cohorts including a febrile rash cohort (attempting to capture acute Zika/Chikungunya/Dengue infection), a household cohort (attempting to capture asymptomatic or minimally symptomatic subjects), and a cohort of those with Guillain Barré). Additionally, two subpopulations of the febrile rash cohort that have special follow up. This includes the pregnant population, who will be followed through delivery to determine pregnancy outcomes, and those subjects with neurologic or cognitive manifestations who will be evaluated to determine the spectrum of neurologic disease seen with these diseases.

Subjects with Guillain Barré with potential exposure to Zika virus are of special interest given the severity of disease. Subjects with Guillian Barré do not need to have a preceding illness suggestive of Zika or other viruses. As there are few subjects with Guillain Barré, subjects will be enrolled in two ways - a prospective cohort for subjects with acute Guillain Barré, and a cohort for subjects that had Guillain Barré in the last several years. Data collected systematically from these cohorts will improve the understanding of Zika/Chikungunya/Dengue virus infections.

There are many uncertainties about the number of subjects that meet this case definition. There are limits to the ability to enroll based on staffing and other resources. If there are many cases, an emphasis will be placed on enrolling pregnant subjects and adults with neurologic complications that meet the case definition, as this is the area of highest clinical need. If there are few pregnant women or subjects with neurologic problems that can be enrolled, then any adults or children meeting the criteria can be enrolled. Not all cohorts will be active at all sites, based on the type of facility and type of patients typically seen. If sufficient numbers of certain populations are enrolled (i.e. children born to women infected with Zika), the protocol may be amended to study those populations in more detail.

ELIGIBILITY:
Febrile Rash Cohort Inclusion Criteria:

Subjects with fever and/or rash will be included if they are 1 year of age or older, and meet one of the following criteria (1 or 2):

1. Meeting the WHO/PAHO case definition, as defined as (a and b and c):

   1. One or both of the following primary signs:

      * Rash
      * Elevated body temperature (> 37.2 °C) AND
   2. One or more of the following symptoms (not explained by other medical conditions):

      * Arthralgia
      * Myalgia
      * Non-purulent conjunctivitis or conjunctival hyperemia
      * Headache
      * Malaise AND
   3. Onset of illness in the last 7 days
2. Modified case definition (a and b):

   1. Any two of the following:

      * Rash
      * Elevated body temperature (> 37.2 °C)
      * Arthralgia
      * Myalgia
      * Non-purulent conjunctivitis or conjunctival hyperemia
      * Headache
      * Malaise AND
   2. Onset of illness in the last 7 days

Household Cohort Inclusion Criteria:

1. 1 year of age and older, and
2. Either live in the same household as a subject enrolled into the febrile rash cohort OR live in the same household as a subject who is experiencing an illness similar to Zika (fever and rash as previously described), regardless if said subject is enrolled in the study.

Guillain-Barré Prospective Cohort Inclusion Criteria:

Either confirmed or suspected Guillain-Barré (areflexic flaccid paralysis) as defined either of the following:

1. Confirmed Guillain-Barré

   1. Acute onset of weakness or paralysis (from baseline to full weakness in 20 days)
   2. Weakness is symmetrical
   3. Areflexic (reflexes are 0/4)
2. Suspected Guillain-Barré

   1. Acute onset of illness
   2. Areflexic flaccid paralysis

Prior Guillain-Barré Cohort Inclusion Criteria:

1. Confirmed Guillain-Barré

   1. Acute onset of weakness or paralysis (from baseline to full weakness in 7 days)
   2. Weakness is symmetrical
   3. Areflexic (reflexes are 0/4)
   4. Diagnosis since January 2014
2. Suspected Guillain-Barré

   1. Acute onset of illness
   2. Areflexic flaccid paralysis
   3. Clinical diagnosis of Guillain-Barré
   4. Diagnosis since January 2014

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will recruit male and female individuals of one year of age or older from southeastern Mexico and neighboring areas who exhibit signs of rash and/or fever that may be indicative Zika, Dengue, or Chikungunya. In addition, family members of these individuals will asked to be participate whether they have symptoms or not. Pregnant women will be included. Also, all individuals with a prior diagnosis of Guillain-Barré or history suggestive of Guillain-Barré will be asked to enroll.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects that have confirmed Zika, Chikungunya, or Dengue (including co-infections) from the subjects presenting with fever and/or rash in southeastern Mexico. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Siddiqui, Study Chair — National Institute of Allergy and Infectious Diseases (NIAID); Guillermo Ruiz-Palacios, Study Chair — Mexican Emerging Infectious Diseases Clinical Research Network; Pablo Francisco Belaunzarán Zamudio, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (6):
- Mexico (6):
  - Hospital General de Tapachula, Tapachula, Chiapas
  - Hospital Regional de Alta Especialidad Ciudad Salud, Chiapas
  - Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (ISSSTE) Clínica Hospital Dr. Roberto Nettel Flores, Chiapas
  - Instituto Mexicano del Seguro Social (IMSS) Delegación Estatal / Hospital General de Zona con Medicina Familiar No. 1, Chiapas
  - Instituto Mexicano del Seguro Social (IMSS) Delegación Estatal / Unidad de Medicina Familiar No. 11, Chiapas
  - Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belaunzaran-Zamudio PF, Rincon Leon HA, Caballero Sosa S, Ruiz E, Najera Cancino JG, de La Rosa PR, Guerrero Almeida ML, Powers JH 3rd, Beigel JH, Hunsberger S, Trujillo K, Ramos P, Arteaga-Cabello FJ, Lopez-Roblero A, Valdes-Salgado R, Arroyo-Figueroa H, Becerril E, Ruiz-Palacios G; Mexican Emerging Infectious Diseases Clinical Research Network (La Red). Different epidemiological profiles in patients with Zika and dengue infection in Tapachula, Chiapas in Mexico (2016-2018): an observational, prospective cohort study. BMC Infect Dis. 2021 Aug 28;21(1):881. doi: 10.1186/s12879-021-06520-x. PMID 34454432
- [Derived] Belaunzaran-Zamudio PF, Ortega-Villa AM, Mimenza-Alvarado AJ, Guerra-De-Blas PDC, Aguilar-Navarro SG, Sepulveda-Delgado J, Hunsberger S, Salgado RV, Ramos-Castaneda J, Rincon Leon HA, Rodriguez de La Rosa P, Najera Cancino JG, Beigel J, Caballero Sosa S, Ruiz Hernandez E, Powers JH 3rd, Ruiz-Palacios GM, Lane C. Comparison of the Impact of Zika and Dengue Virus Infection, and Other Acute Illnesses of Unidentified Origin on Cognitive Functions in a Prospective Cohort in Chiapas Mexico. Front Neurol. 2021 Mar 22;12:631801. doi: 10.3389/fneur.2021.631801. eCollection 2021. PMID 33828518
- [Derived] Gouel-Cheron A, Lumbard K, Hunsberger S, Arteaga-Cabello FJ, Beigel J, Belaunzaran-Zamudio PF, Caballero-Sosa S, Escobedo-Lopez K, Ibarra-Gonzalez V, Najera-Cancino JG, Rincon-Leon HA, Ruiz-Hernandez E, Sepulveda-Delgado J, Trujillo-Murillo K, Ruiz-Palacios G. Serial real-time RT-PCR and serology measurements substantially improve Zika and Dengue virus infection classification in a co-circulation area. Antiviral Res. 2019 Dec;172:104638. doi: 10.1016/j.antiviral.2019.104638. Epub 2019 Oct 28. PMID 31672665